CLINICAL TRIAL: NCT05117528
Title: Streptococcus Pyogenes Carriage Acquisition, Persistence and Transmission Dynamics Within Households in The Gambia: a Longitudinal Cohort Study
Brief Title: Streptococcus Pyogenes Carriage Acquisition and Transmission Study
Acronym: SpyCATS
Status: Completed | Type: Observational
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Other Study IDs: LEO 24005
Record Dates: First submitted 2021-04-21; First posted 2021-11-11 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Group A Streptococcal Infection; Scabies; Microbial Colonization
Keywords: Group A Streptococcal skin colonization; Group A Streptococcal pharyngeal carriage; Group A Streptococcal transmission
MeSH Terms: conditions — Streptococcal Infections; Scabies; Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Oropharyngeal swabs Normal skin swabs Pyoderma wound swabs Blood Serum Dried Blood Spot Oral fluid Environmental swabs Settle plates
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Group A Streptococcus (GAS) is a bacteria which causes severe infections and leads to deadly diseases such as rheumatic heart disease which kills over 300,000 people a year globally, particularly in low-income countries. It is not know how GAS is spread between people, how often people carry GAS in their throat or on their skin without having symptoms, or what factors increase the chance of this occurring. It is important to understand these factors in order to know how to reduce GAS-related disease.

This study will follow 444 people in The Gambia, over 12 months, taking samples from the throats and skin of people living in the same households, and asking questions about themselves and their behaviour, at regular intervals. By taking samples over time, the investigators hope to understand how common it is to carry GAS without having symptoms, how GAS is spread between people, and whether carrying GAS leads to more GAS infections in people or their household members.

The study will use state-of-the-art techniques to look at the DNA of GAS bacteria that we find, and combine this with a mathematical model to investigate how different strains spread to people within and between households in the community.

DETAILED DESCRIPTION:
Type of study and design

The study is a prospective, longitudinal (open) cohort study within households in Sukuta, The Gambia. Households will be recruited, and all available household members asked to participate. Households will be followed for 12 months, with up to monthly visits (at least 3-monthly visits), and more frequently for some subgroups of participants.

A total of 45 households will be recruited, including every available household member as individual participants (resulting in a cohort of approximately 450 participant with the average household size in Sukuta being around 10).

Households will be enrolled for 12 months, with enrolment aiming to commence before the rainy season, to ensure that the enrolment period will span one full rainy season, with dry periods either side. Every household will undergo an enrolment visit (MV0), then up to monthly visits (MV1, MV2, MV3 etc., up to MV12) or less frequently if practical constraints arise.

At each visit an oropharyngeal swab, normal skin swab, oral fluid sample and dried blood spot sample will be taken from all individuals, data collected on socio-demographics, social mixing behaviour and clinical examination findings. Examination findings recorded will include evidence of pharyngitis, pyoderma, and scabies. In addition, a blood sample for serum will be taken at the beginning and end of the study for detailed functional immune responses. Swabs will also be taken from any pyoderma lesions, from common touch points in the household such as door handles, and settle plates used inside households.

Swabs will be transported the same day to the laboratory and plated for microbiological culture. The culture will identify the presence of GAS from the swabs, and if present, antibiotic resistance will be determined and isolates stored for later use. Additionally, if Groups C and G Streptococcus are identified the isolates will be stored, and from normal skin and pyoderma wound swabs, any Staphylococcus aureus isolates will stored.

Swabs from participants will be cultured for the presence of GAS and isolates will undergo whole genome sequencing in order to assess phylogenetic relatedness of strains identified. These data, combined with temporal incidence of strain acquisition, clinical data and household situation will be used to build a mathematical model of GAS transmission to identify key routes of transmission within and between households.

Sub-studies:

Intensified incident GAS surveillance cohort

A subgroup of 12 households, most with at least one asymptomatic GAS carrying individual at baseline, and some with no carriers, will form a cohort to undergo intensified swabbing. This cohort will be used to assess incidence of GAS carriage and disease with greater resolution than the main cohort. All household members present will undergo more frequent swabbing, with a view to being visited every week for 6 months. At these visits, more detailed social-mixing behaviour data will be collected.

Estimating duration of GAS carriage

A further subgroup will also be identified to allow for greater resolution in the estimation of the duration of GAS carriage. Following enrolment, any participant who becomes GAS carrier positive (i.e. was negative at baseline or the previous visit, and then becomes positive asymptomatically) will have weekly swabs taken from the same site that was positive, until 2 GAS negative swabs have been taken in a row.

Estimating GAS infection incidence

To assess incidence of clinical GAS disease in the cohort throughout the study, all participants reporting symptoms suggestive of possible clinical GAS infection such as pharyngitis or pyoderma (but also including invasive infections), will be visited for an unscheduled visit where a clinical and health-seeking history will be recorded, a swab, saliva and DBS taken, and treatment (or further management) will be delivered according to WHO guidelines or best local practice. Furthermore, at each scheduled visit, any individual identified with symptoms of clinical GAS infection will undergo the same process of history-taking, swabbing, treatment and follow up.

ELIGIBILITY:
Inclusion Criteria:

Households must:

* Be within the boundary of Sukuta as determined by the 2013 census
* Have at least 3 members including at least one child under age 18

Individuals must:

* Provide signed (or thumbprinted) informed consent for study participation (obtained from a parent or guardian for children under the age of 18
* Be willing and have capacity to participate and comply with the study protocol as judged by a member of the study team
* Be resident in the household, with no plans to move outside of the household during the period of study participation

Exclusion Criteria:

Households:

- Less than 80% of individuals living in the household, as defined by the The Gambia Demographic and Health Survey 2013 definition, provide consent to participate

Individuals:

* Consent not provided
* Has any condition or any other reason that may lead to difficulty or discomfort in obtaining all the necessary samples
* Is judged by the study team member to be unable or unlikely to participate and comply with the study protocol for the entire study period

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Sukuta is an area within the West Coast Region peri-urban conurbation of The Gambia, with a population of 47,048 in 2013, including 7,234 children aged under 5 years, and an average household size of 8.1. The Gambia is the smallest mainland country in Africa with a population of 1.9 million in 2013 and was ranked 174th in the world in the UN Human Development Index in 2017.
  Households within the 2013 boundaries of Sukuta will be randomly selected using a list of randomly generated GPS locations stratified by housing density (high, medium and low). All eligible and willing households identified using the GPS location list will be enrolled, until the target sample size of 45 households is reached.
  All individuals living within the households will be enrolled, with no age restrictions.
Sampling Method: Probability Sample
Enrollment: 441 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of oropharyngeal swabs positive for GAS each month | Monthly visits
  Oropharyngeal swabs taken at monthly visits will be plated for microbiological culture, and the presence of GAS determined by latex agglutination testing.
Prevalence of normal skin swabs positive for GAS each month | Monthly visits
  Normal skin swabs taken at monthly visits will be plated for microbiological culture, and the presence of GAS determined by latex agglutination testing.
Incidence of GAS-positive oropharyngeal swabs | 1 year
  Oropharyngeal swabs taken at each visit will be plated for microbiological culture, and the presence of GAS determined by latex agglutination testing. The incidence of positive swabs in person-years will be calculated
Incidence of GAS-positive normal skin swabs | 1 year
  Normal skin swabs taken at each visit will be plated for microbiological culture, and the presence of GAS determined by latex agglutination testing. The incidence of positive swabs in person-years will be calculated
Change in GAS-positive swabs per month | 1 year
  Seasonal changes in GAS-positivity will be assessed over the course of a year.

SECONDARY OUTCOMES:
Adjusted hazard ratio for GAS carriage depending on presence of relevant risk factors | 1 year
Adjusted hazard ratio for GAS symptomatic infection depending on presence of relevant risk factors | 1 year
Difference in GAS emm type diversity compared to other settings | 1 year
The level of GAS tissue tropism | 1 year
Prevalence of Group C streptococcal carriage | Monthly
Prevalence of Group G streptococcal carriage | Monthly
Prevalence of Staphylococcus aureus skin carriage | Monthly
Seroprevalence of anti-GAS antibodies | Baseline
Sensitivity of GAS isolates to antimicrobials. | 1 year
Difference in GAS-specific serological immune activity between GAS-colonised and non-GAS colonised participants | 1 year
Difference in GAS-specific mucosal immune activity between GAS-colonised and non-GAS colonised participants | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Edwin P Armitage, BMBS, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- MRC Unit The Gambia at LSHTM, Fajara, The Gambia

IPD SHARING:
Plan to Share IPD: Yes
Anonymised raw data for all analysis performed during manuscript preparation will be published alongside the manuscripts. All other data will be archived at the MRC Unit The Gambia and will be made available to other researchers upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data used for manuscript preparation will be made available at the time of publication for as long as the journal makes it available.

REFERENCES:
- [Derived] de Crombrugghe G, Armitage EP, Keeley AJ, Senghore E, Camara F, Jammeh M, Bittaye A, Ceesay H, Ceesay I, Samateh B, Manneh M, Botquin G, Lakhloufi D, Delforge V, Bah SY, Hall JN, Schiavolin L, Turner CE, Marks M, de Silva TI, Botteaux A, Smeesters PR; MRCG StrepA Study Group. Household Molecular Epidemiology of Streptococcus pyogenes Carriage and Infection in The Gambia. J Infect Dis. 2025 Sep 15;232(3):550-559. doi: 10.1093/infdis/jiaf252. PMID 40378280
- [Derived] Armitage EP, de Crombrugghe G, Keeley AJ, Senghore E, Camara FE, Jammeh M, Bittaye A, Ceesay H, Ceesay I, Samateh B, Manneh M, Kampmann B, Turner CE, Kucharski A, Botteaux A, Smeesters PR, de Silva TI, Marks M; MRCG StrepA Study Group. Streptococcus pyogenes carriage and infection within households in The Gambia: a longitudinal cohort study. Lancet Microbe. 2024 Jul;5(7):679-688. doi: 10.1016/S2666-5247(24)00046-6. Epub 2024 May 9. PMID 38735305

DOCUMENTS (1):
  • Study Protocol (2022-04-18): https://cdn.clinicaltrials.gov/large-docs/28/NCT05117528/Prot_000.pdf